CLINICAL TRIAL: NCT06566612
Title: Avoidance-driven Decision Making and Learning in Anorexia Nervosa and Bulimia Nervosa
Status: Recruiting | Type: Observational
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Christina Wierenga, Professor in Residence, University of California, San Diego
Other Study IDs: 810384
Record Dates: First submitted 2024-08-15; First posted 2024-08-22 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Bulimia Nervosa; Anorexia Nervosa
MeSH Terms: conditions — Bulimia Nervosa; Anorexia Nervosa

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Anorexia Nervosa: Participants that meet Diagnostic And Statistical Manual Of Mental Disorders (DSM-V) criteria for Anorexia Nervosa.
- Bulimia Nervosa: Participants that meet DSM-V criteria for Bulimia Nervosa.
- Healthy Controls: Participants that do not meet DSM-V criteria for any disorder.

SUMMARY:
The purpose of this study is to investigate areas of the brain responsible for avoidance learning in adults with eating disorders using brain imaging techniques, computer tasks, and self-report questionnaires and interviews. The investigators will study changes in brain activity using a procedure called functional magnetic resonance imaging (fMRI). This study will include 78 women with an eating disorder (26 with anorexia nervosa [AN], 26 with bulimia nervosa [BN]) and 26 healthy controls (HC) aged 18-39.

Aim 1: Evaluate behavioral differences in active and passive avoidance learning in eating disorders and associations with symptoms.

Aim 2: Evaluate whether corticostriatal and limbic-prefrontal fMRI BOLD response associated with avoidance learning differs in eating disorders relative to healthy controls and relates to symptoms.

Aim 3: Evaluate whether functional connectivity of avoidance learning neural circuity differs in eating disorders relative to healthy controls.

ELIGIBILITY:
Inclusion Criteria:

Eating Disorder Group:

* Between the ages of 18 and 39 years old
* Meet DSM-V criteria for anorexia nervosa or bulimia nervosa

Healthy Controls:

* Between the ages of 18 and 39 years old
* Have maintained 85% to 120% ideal body weight since menarche

Exclusion Criteria:

* Psychotic illness/other mental illness requiring hospitalization
* Current dependence on drugs or alcohol defined by DSM IV criteria. Additionally, positive test results for drug use on the day of the scan, apart of marijuana, will result in cancelling or rescheduling the scan because acute use will impact MRI measures.
* Physical conditions (e.g. diabetes mellitus, pregnancy) known to influence eating or weight
* Neurological disorder, neurodevelopmental disorder, or history of head injury with >30 min loss of consciousness
* Any contraindication to undergoing an MRI
* Primary obsessive compulsive disorder or primary major depressive disorder

Additional Exclusion Criteria for ED Group:

* If taking other psychotropic medication, any change in dosage in the 2 weeks before scanning

Additional Exclusion Criteria for Healthy Control Group:

* Meet criteria for the diagnosis of any psychiatric disorder currently
* Any history of binge eating or purging behaviors, including self-induced vomiting, laxative or diuretic misuse
* Use of any psychoactive or other medication known to affect mood or concentration in the last 3 months

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study will recruit 52 adult women currently ill with an eating disorder, including anorexia nervosa (AN; n=26) and bulimia nervosa (BN, n=26), and 26 healthy control (HC) women between the ages of 18 and 39.
Sampling Method: Non-Probability Sample
Enrollment: 78 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Learning rate | 25 minutes
  Behavioral responses during a card game gambling task
fMRI brain response | 25 minutes
  fMRI brain activity associated with the card game gambling task
Brain connectivity | 10 minutes
  Whole-brain functional connectivity associated with the card game gambling task

CONTACTS AND LOCATIONS:
Locations (1):
- UCSD Eating Disorders Treatment and Research Program, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: Undecided